CLINICAL TRIAL: NCT06747104
Title: Assessment of Upper Limb Muscle Activity and the Effect of Manual Therapy on Fatigue, Stiffness and Muscle Activity During Training
Brief Title: Application of Manual Therapy to Archers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KB/750/2023-2024
Record Dates: First submitted 2024-12-08; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: archery; muscle fatigue; recovery; manipulation
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assessment of acute effects of manipulation and muscle strength (Active Comparator): Performing the manipulation with a preliminary two-second tension of the joint capsule in the shoulder and elbow joints.
  Interventions: Other: Manual therapy; Other: Placebo

INTERVENTIONS:
Other: Manual therapy — This technique involves a low-amplitude, high-velocity push on the shoulder and elbow joints with an additional two-second tension
Other: Placebo — Performing manipulations without a two-second preliminary tension of the joint capsule in the shoulder and elbow joints.

SUMMARY:
The aim of this study is to: (i) characterize the effect of repeated archery shots on the EMG parameters of certain selected upper limb muscles; and (ii) evaluate how manipulation of the initial two-second tension phase, in particular involving muscle stretching, affects these EMG parameters after repeated shots.

DETAILED DESCRIPTION:
EMG measurements will be collected for selected muscles in the shoulder joint and forearm, at points: initially at the beginning, after the athletes have performed 50 and another 50 archery shots, and finally after undergoing manual therapy. The main phase of muscle testing will take place in the Aiming phase.

ELIGIBILITY:
Inclusion Criteria:

* Actively training as an archer at least twice a week for six months;
* In good health, with no recent injury or illness;
* Over 18 years of age;
* Engagement in all phases of the study.

Exclusion Criteria:

* Any injury or illness present at the time of the study;
* Recent history (within six months) of upper extremity injury (shoulder, elbow, or wrist), joint pain, lower extremity joint hypermobility, or neurological/connective tissue disease.
* No training participation
* No consent for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of MVC. | Each isometric muscle test lasts 3 seconds. The study is performed three times for each muscle.
  Muscle EMG is an assessment of the electrical characteristics during the study, the electrical source of which is the muscle membrane potential, and the measured EMG potentials are measured in μV and the repetition rate of muscle motor unit firing measured in Hz, at the same time of the study.
Muscle stiffness | Each Myoton application lasts 1 sec for one point. Three evaluations of one of the two points for one muscle are performed. It is assumed that the study with recording will last 30 seconds for one muscle.
  Muscle stiffness - characteristic resistance to physical contraction, which deforms initially forming. Stiffness (N/m) was calculated as S = amax.mprobe/Δl.

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Studnicki, PhD, Principal Investigator — Medical University of Gdansk

IPD SHARING:
Plan to Share IPD: No
Once the study is complete, the results will be sent to the researcher who will analyze the data.